CLINICAL TRIAL: NCT03633149
Title: Tablet-based Intervention to Prevent Substance-exposed Pregnancy in Primary Care
Brief Title: Choices4Health: Intervention to Prevent Substance-exposed Pregnancy
Acronym: C4H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Baylor College of Medicine (Other); The University of Texas Health Science Center, Houston (Other); University of Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01AA022924 (NIH)
Record Dates: First submitted 2016-05-11; First posted 2018-08-16 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Prenatal Alcohol Exposure; Prenatal Tobacco Exposure; Prenatal Marijuana Exposure
Keywords: prenatal alcohol exposure; marijuana; smoking cessation; computer-delivered intervention; contraception; behavioral intervention; motivational interviewing
MeSH Terms: conditions — Marijuana Abuse; Smoking Cessation | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Computer tablet-delivered C4H (Experimental): Two session CHOICES4Health intervention delivered by a computer tablet to address no use or ineffective use of contraception, and risky alcohol use, or cigarette smoking, or marijuana use.
  Interventions: Behavioral: Computer tablet-delivered C4H
- Person-delivered C4H (Experimental): Two session CHOICES4Health intervention delivered by a counselor to address no use or ineffective use of contraception, and risky alcohol use, or cigarette smoking, or marijuana use.
  Interventions: Behavioral: Person-delivered C4H
- Brief Advice (Active Comparator): Women will receive advice and educational material from a research assistant about risk drinking, smoking, marijuana, and contraception, depending on their specific risk behaviors, as well as information about women's health. In addition, the women will receive referrals to the Harris Health System's SBIRT clinic if needed.
  Interventions: Behavioral: Brief Advice

INTERVENTIONS:
Behavioral: Computer tablet-delivered C4H — Two session CHOICES intervention targeting ineffective contraception and risky alcohol use and/or cigarette smoking and/or marijuana use to reduce the risk of a substance-exposed pregnancy delivered on a computer-tablet.
  Other Names: C4H-T
  Arms: Computer tablet-delivered C4H
Behavioral: Person-delivered C4H — Two session CHOICES intervention targeting ineffective contraception and risky alcohol use and/or cigarette smoking and/or marijuana use to reduce the risk of a substance-exposed pregnancy delivered by a counselor.
  Other Names: C4H-C
  Arms: Person-delivered C4H
Behavioral: Brief Advice — Brief advice delivered by a research associate about healthy behaviors for women including use of contraception and alcohol, tobacco, and marijuana use
  Other Names: BA
  Arms: Brief Advice

SUMMARY:
This is a 4-year randomized, controlled study to test the efficacy of the CHOICES4Health-T (C4H-T) delivered by a computerized tablet, CHOICES4Health-C (C4H-C), delivered by a counselor, and brief advice (BA), on reducing preconception substance-exposed pregnancy risk (i.e. drinking below risk levels; tobacco and marijuana cessation; effective contraception use) among women (aged 18-44) presenting to the 13 primary care clinics that serve adults within the Harris Health System. Given the natural fit between contraceptive and HIV prevention counseling the CHOICES4Health interventions will also target HIV sexual risk behaviors.

DETAILED DESCRIPTION:
A randomized group design (N = 240) will be used to test the efficacy of the C4H-C and C4H-T interventions relative to Brief Advice (BA) to reduce the risk of substance-exposed pregnancy) SEP in preconception women of childbearing age. Follow-up assessments will be conducted at 3, 6, and 9 months.

Each of the substances targeted in this study (risk drinking, cigarette smoking, and marijuana use) is commonly used relative to other substances and is singly or jointly associated with risk for poor fetal outcomes. Thus, women who are not using effective contraception (i.e., use of effective birth-control methods during all vaginal intercourse) and have any one or more substance-risk behaviors in the 30 days before intake will be eligible for the study.

Urn randomization will be used to stratify women on all three substance-risk behaviors to ensure a balanced number of women presenting with alcohol-exposed pregnancy (AEP), tobacco-exposed pregnancy (TEP), and marijuana-exposed pregnancy (MEP) risks across the three study conditions. To address risk distribution for women who present with more than one risk behavior the urn randomization will also be programmed to balance single risk and multiple risk women across the study conditions. In sum, the urn randomization will include four assignment criteria: AEP, TEP, MEP, and multiple risks. Finally, different numbers of women will be needed for each type of substance-exposed pregnancy risk in order to provide sufficient power for the investigator's analytic tests. For example, approximately 25% more women at risk of AEP are required than for TEP to attain the same power. The investigators will include over sampling rules and stopping rules to ensure adequate recruitment for AEP, TEP, and MEP.

ELIGIBILITY:
Inclusion Criteria: Women who:

* are 18-44 years old;
* have no condition causing infertility (e.g., tubal ligation, hysterectomy, menopause);
* are not pregnant or planning to become pregnant in the next 12 months;
* are available for the follow-up period;
* had vaginal intercourse during the previous 30 days with a fertile man and did not use effective contraception every time AND are drinking at risk levels (more than 3 drinks/day or more than 7 drinks/week); OR are reporting marijuana use in the previous month, OR are currently smoking cigarettes (at least weekly use) during the 30-day baseline period.

Exclusion Criteria: Women who:

* have severe cognitive, and/or psychiatric impairment that precludes cooperation with study protocol, per judgment of the C4H interventionist or research staff;
* are unable to read, write, and speak English or Spanish;
* are unable or unwilling to meet study requirements, including followup assessments.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 219 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in risk of alcohol-exposed pregnancy (AEP) as measured by self-reported daily standard drinks, vaginal sex, and use of contraception on the Timeline Followback calendar. | 3, 6, and 9 months
  Risk of AEP is defined as any risk drinking (>3 drinks/day or >7 drinks/week on average) and any occurrence of vaginal sex with no use or ineffective use of contraception in the assessment period. Self-reported daily alcohol use (in standard drinks), vaginal intercourse, and contraception (effective use) data from the Timeline Followback will be used to calculate risk of AEP for the previous 90 days. Change in Risk of AEP will be examined at 3-, 6-, and 9-months post-intake. A participant will be considered at risk of AEP at each of the 3-, 6-, and 9 month timepoints if the participant had any occurrence of vaginal sex without the use of effective contraception and had more than 3 standard drinks on any day or more than 7 standard drinks per week on average in any 30 day period in the previous 90 days. Risk of AEP will be a dichotomous outcome (at risk of AEP or at reduced risk of AEP).
Change in risk of tobacco-exposed pregnancy (TEP) as measured by self-reported daily number of cigarettes, vaginal sex, and use of contraception on the Timeline Followback calendar. | 3, 6, and 9 months
  Risk of TEP is defined as currently smoking cigarettes (at least weekly use) and any occurrence of vaginal sex with no use or ineffective use of contraception in the assessment period. Self-reported data from the Timeline Followback will be used to calculate risk of TEP for the previous 90 days at 3-, 6 , and 9 months post-intake. A participant will be considered at risk of TEP at each of the 3-, 6-, and 9 month timepoints if the participant had any occurrence of vaginal sex without the use of effective contraception and she had at least weekly smoking in any 30 day period in the previous 90 days. Risk of TEP will be a dichotomous outcome (at risk of TEP or at reduced risk of TEP).
Change in risk of marijuana-exposed pregnancy (MEP) as measured by self-reported marijuana use, vaginal sex, and use of contraception on the Timeline Followback calendar. | 3, 6, and 9 months
  Risk of MEP is defined as any day with marijuana use and any occurrence of vaginal sex with no use or ineffective use of contraception in the assessment period. Self-reported data from the Timeline Followback will be used to calculate risk of MEP for the previous 90 days at 3-, 6- , and 9 months post-intake. A participant will be considered at risk of MEP at each of the 3-, 6-, and 9 month timepoints if the participant had any occurrence of vaginal sex without the use of effective contraception and had any day with marijuana use in any 30 day period in the previous 90 days. Risk of MEP will be a dichotomous outcome (at risk of MEP or at reduced risk of MEP).
Change in risk drinking as measured by self-reported number of standard drinks on the Timeline Followback calendar. | 3, 6, and 9 months
  Risk drinking is defined as drinking more than 3 standard drinks on any day or drinking more than 7 standard drinks in a week on average in the previous 90 days. Self-reported data from the Timeline Followback will be used to calculate risk drinking for the previous 90 days at 3-, 6-, and 9-months post-intake. Risk drinking will be a dichotomous outcome (yes or no).
Change in cigarette smoking as measured by self-reported number of cigarettes smoked each day on the Timeline Followback calendar. | 3, 6, and 9 months
  Cigarette smoking is defined as at least weekly cigarette smoking in the previous 90 days on the Timeline Followback calendar at 3-, 6-, and 9-months post-intake. Cigarette smoking will be a dichotomous outcome (yes or no). In addition, smoking will be validated using biological test to assess cotinine levels.
Change in marijuana use as measured by self-reported use for each day on the Timeline Followback calendar. | 3, 6, and 9 months
  Marijuana use is defined as any day with any marijuana use in the previous 90 days on the Timeline Followback calendar at 3-, 6-, and 9-months post-intake. Marijuana use will be a dichotomous outcome (yes or no). In addition, marijuana use will be validated using a biological test to assess Tetrahydrocannabinol (THC) levels.

CONTACTS AND LOCATIONS:
Overall Officials: Mary M Velasquez, Ph.D., Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Health Behavior Research and Training Institute, University of Texas at Austin — https://sites.utexas.edu/hbrt/

DOCUMENTS (1):
  • Informed Consent Form (2019-08-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT03633149/ICF_000.pdf